CLINICAL TRIAL: NCT06162299
Title: A Phase I, Double-blind, Randomized, Placebo-controlled, Dose Escalating Study to Evaluate the Safety, Immunogenicity and Efficacy of YS-HBV-002 in the Treatment of Chronic Hepatitis B (CHB) Infection in Adults ≥ 18 Years Old
Brief Title: A Phase I, the Study to Evaluate the Safety, Immunogenicity and Efficacy of YS-HBV-002
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business strategy
Sponsor: Yisheng Biopharma (Singapore) Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YS-101
Record Dates: First submitted 2023-11-22; First posted 2023-12-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Chronic Hepatitis B
Keywords: PIKA Adjuvant
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose 0.5mL (Experimental): Group A ：The first 4 enrollees in Group A will be sentinel patients and will be allocated at a 1:1 ratio to receive 0.5mL of either YS-HBV-002 or placebo(saline solution), The next 12 enrollees in Group A will be the main patients and will be allocated at 5:1 to receive 0.5mL of either YS-HBV-002 or placebo.
  Interventions: Biological: YS-HBV-002
- Mid-dose 1.0mL (Experimental): Group B ：The first 4 enrollees in Group B will be sentinel patients and will be allocated at a 1:1 ratio to receive 1.0mL of either YS-HBV-002 or placebo(saline solution), The next 12 enrollees in Group A will be the main patients and will be allocated at 5:1 to receive 1.0mL of either YS-HBV-002 or placebo.
  Interventions: Biological: YS-HBV-002
- High dose 2.0mL (Experimental): Group C ：The first 4 enrollees in Group C will be sentinel patients and will be allocated at a 1:1 ratio to receive 2.0mL of either YS-HBV-002 or placebo(saline solution), The next 12 enrollees in Group A will be the main patients and will be allocated at 5:1 to receive 2.0mL of either YS-HBV-002 or placebo.
  Interventions: Biological: YS-HBV-002

INTERVENTIONS:
Biological: YS-HBV-002 — YS-HBV-002, A recombinant hepatitis B vaccine with PIKA adjuvant

SUMMARY:
This is the first-in-human Phase I, double-blind, randomized, placebo-controlled, dose escalating study to evaluate the safety, immunogenicity and preliminary efficacy of the YSHBV-002 in the treatment of CHB in adults ≥18 years old. There will be 3 escalating doses of YS-HBV-002 to be administered intramuscularly: 0.5mL, 1.0mL, and 2.0mL.

DETAILED DESCRIPTION:
This is the first-in-human Phase I, double-blind, randomized, placebo-controlled, dose escalating study to evaluate the safety, immunogenicity and preliminary efficacy of the YSHBV-002 in the treatment of CHB in adults ≥18 years old. There will be 3 escalating doses of YS-HBV-002 to be administered intramuscularly: 0.5mL, 1.0mL, and 2.0mL. Enrollment in the study will sequentially start from the low dose 0.5mL as Group A, then to the mid-dose 1.0mL as Group B and lastly to the high dose of 2.0mL as Group C. Each group will have 16 patients enrolled. The first 4 enrollees in Group A will be sentinel patients and will be allocated at a 1:1 ratio to receive 0.5mL of either YS-HBV-002 or placebo (Table 3). As there is no comparable equivalent to YS-HBV-002 available in the market, the placebo of normal saline solution to be injected intramuscularly will serve as the control in this trial. The next 12 enrollees in Group A will be the main patients and will be allocated at 5:1 to receive 0.5mL of either YS-HBV-002 or placebo. The vaccination regimen will be 1 IM injection every 3 days in the deltoid muscle, alternately for approximately 6 weeks. A total of 14 injections will be administered to each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years during screening
2. Body Mass Index (BMI) of 18.5-30 kg/m2
3. Diagnosed or laboratory confirmed to have CHB

   1. Have CHB infection for at least 6 months
   2. HBsAg titer ≥ 1000 IU/mL
   3. HBV DNA ≥ 2000 IU/mL
   4. Serum alanine amino transferase (ALT) and aspartate aminotransferase (AST) ≤ 2 × upper limit of normal (ULN)
4. Able to provide informed consent
5. Able and willing to comply with all study procedures throughout the study period of approximately 3 months
6. For female subjects with childbearing potential: must agree to avoid pregnancy throughout the study period of approximately 3 months. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods on avoiding pregnancy include: a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with a spermicide.

Exclusion Criteria:

1. Pregnant or breastfeeding or intending to become pregnant within the projected duration of the trial
2. Transient elastography at screening revealing a FibroScan value of ≥ 9 kPa or a previous liver biopsy evidencing hepatic fibrosis at or within 24 months prior to vaccination
3. Patients with hepatitis caused by other etiologies
4. History of or manifestations of liver decompensation (e.g., Child-Pugh Class B or C, or ascites, gastrointestinal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis, etc....)
5. Currently participating in or has participated in a study with an IP within 30 days preceding Day 0
6. Fever (axillary temperature ≥ 37.8 ℃)
7. Subjects with abnormal indicators of blood biochemistry and other routine blood tests deemed clinically significant by the investigator
8. History of severe allergic reactions (such as acute anaphylaxis, urticaria, skin eczema, dyspnea, angioneurotic edema, or allergic abdominal pain) or allergy to any of the components of YS-HBV-002
9. Any history of anaphylaxis or angioedema after any vaccination
10. Allergy to kanamycin and aminoglycosides
11. Past or family history of convulsion, epilepsy, encephalopathy, or mental illness
12. Diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia, or other autoimmune diseases
13. History of coagulation dysfunction (e.g., coagulation factor deficiency, coagulation disease)
14. Bleeding disorder, or receipt of anticoagulants in the past 21 days preceding inclusion, contraindicating IM vaccination based on the investigator's judgement
15. Vaccinated with live attenuated vaccine within 1 month, or other vaccine/non-COVID-19 vaccine within 14 days prior to vaccination
16. Receiving immunotherapy or inhibitor therapy (consistently oral or infusion for more than 14 days) within 3 months prior to vaccination
17. Received systemic immunosuppressants within 4 months prior to vaccination or anticipating the need for immunosuppressant at any time during participation in the study. Topical or inhaled treatment is allowed if not used within 14 days prior to vaccination
18. Have received antiviral therapy for chronic hepatitis but have stopped for less than 30 days or plan to take antiviral therapy during the study
19. Received blood products within 3 months before vaccine administration
20. History of alcohol or drug abuse within the past 2 years
21. Any condition that, in the opinion of the investigator, would pose a health risk to the patient if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs within 30 minutes after vaccination. | 30 minutes post each vaccination
  To assess the safety and tolerability
Incidence of solicited local reactions within 7 days after each vaccination. | 7 days post each vaccination
  To assess the safety and tolerability
Incidence of solicited systemic reactions from first vaccination to 7 days after the last vaccination (D1 to D46). | From Day1 to Day46
  To assess the safety and tolerability
Incidence of unsolicited AEs, serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs), adverse events of special interest (AESIs), and AEs leading to withdrawals throughout the study period | From Day1 to Day 90
  To assess the safety and tolerability

SECONDARY OUTCOMES:
Proportion of patients showing reduction in HBV DNA using PCR for each dose from baseline to the end of the study and at specified timepoints. | Day0， Day16， Day34， Day60， Day90
  To evaluate the preliminary efficacy, immunogenicity and determine the appropriate dose
Change in mean log10 of HBV DNA from baseline to end of study and at each specified timepoint. | Day0， Day16， Day34， Day60， Day90
  To evaluate the preliminary efficacy, immunogenicity and determine the appropriate dose
Change in serum levels of HBeAg, HBcAg, and HBsAg from baseline to end of study at each specified timepoint. | Day0， Day16， Day34， Day60， Day90
  To evaluate the preliminary efficacy, immunogenicity and determine the appropriate dose
Change in serum levels of HBeAg, HBcAg, and HBsAg from baseline to end of study and at each specified timepoint. | Day0， Day16， Day34， Day60， Day90
  To evaluate the preliminary efficacy, immunogenicity and determine the appropriate dose
Proportion of patients with loss (defined as lower limit of quantitation [LLOQ]) or decline in HBsAg, HBcAg, and HBeAg from baseline to the end of the study and at each specified timepoint. | Day0， Day16， Day34， Day60， Day90
  To evaluate the preliminary efficacy, immunogenicity and determine the appropriate dose
GMTs of antibodies against HBsAg, HBcAg and HBeAg at baseline and at pre-defined post-vaccination timepoints. | Day0， Day16， Day34， Day60， Day90
  To evaluate the preliminary efficacy, immunogenicity and determine the appropriate dose
Seroconversion rates of antibodies against HBsAg, HBcAg, and HBeAg. | Day0， Day16， Day34， Day60， Day90
  To evaluate the preliminary efficacy, immunogenicity and determine the appropriate dose

CONTACTS AND LOCATIONS:
Overall Officials: Ike Minerva, MD, Principal Investigator — Iloilo Doctors' Hospiyal
Locations (1):
- Iloilo Doctors' Hospital, Iloilo City, Philippines

IPD SHARING:
Plan to Share IPD: No